CLINICAL TRIAL: NCT06253533
Title: Phase I Clinical Trial on Safety, Tolerability and Immunogenicity of HIV Therapeutic DNA Vaccine (ICVAX) in Clinically Stable HIV Patients Under ART
Brief Title: ICVAX as a HIV Therapeutic DNA Vaccine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immuno Cure Holding (HK) Limited (Industry)
Collaborators: Shenzhen Third People's Hospital (Other); Shenzhen Immuno Cure Biomedical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YKYY-ICVAX-101
Record Dates: First submitted 2024-01-25; First posted 2024-02-12 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Human Immunodeficiency Virus; Human Immunodeficiency Virus I Infection
Keywords: ICVAX; HIV; AIDS; DNA Vaccine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-dose Group (Experimental): Clinically stable HIV-infected patients under ART treatment will receive 1 mg/dose ICVAX or Placebo at 4:1 ratio. ICVAX and Placebo will be administered via intramuscular injection followed by electroporation at 0, 4th, 8th, 12th, and 36th week.
  Interventions: Biological: ICVAX; Other: Placebo
- Medium-dose Group (Experimental): Clinically stable HIV-infected patients under ART treatment will receive 2 mg/dose ICVAX or Placebo at 4:1 ratio. ICVAX and Placebo will be administered via intramuscular injection followed by electroporation at 0, 4th, 8th, 12th, and 36th week.
  Interventions: Biological: ICVAX; Other: Placebo
- High-dose Group (Experimental): Clinically stable HIV-infected patients under ART treatment will receive 4 mg/dose ICVAX or Placebo at 4:1 ratio. ICVAX and Placebo will be administered via intramuscular injection followed by electroporation at 0, 4th, 8th, 12th, and 36th week.
  Interventions: Biological: ICVAX; Other: Placebo

INTERVENTIONS:
Biological: ICVAX — ICVAX is a HIV therapeutic DNA drug developed by Immuno Cure Group based on the PD-1-Enhanced DNA Vaccine Technology platform. The unit dose strength is 2 mg in 1 mL. The dose volume is 0.5 mL/dose for the Low-dose Group, 1.0 mL/dose for the Medium-dose Group, and 2.0 mL/dose for the High-dose Group.
Other: Placebo — Phosphate buffered saline of the same volume will be administered. The dose volume is 0.5 mL/dose for the Low-dose Group, 1.0 mL/dose for the Medium-dose Group, and 2.0 mL/dose for the High-dose Group.

SUMMARY:
The clinical trial is a dose-escalation, randomized, double-blind, placebo-controlled phase I study at a single center to evaluate the safety, tolerability and immunogenicity of HIV Therapeutic DNA Vaccine, ICVAX, in clinically stable HIV patients under ART treatment.

DETAILED DESCRIPTION:
This is a dose-escalation, randomized, double-blind, placebo-controlled phase I study at a single center to evaluate the safety, tolerability and immunogenicity of HIV Therapeutic DNA Vaccine, namely ICVAX, in clinically stable HIV patients under ART treatment. 45 patients will be randomized and divided equally into 3 groups to receive either 1, 2, or 4 mg vaccine or the same volume of placebo at 4:1 ratio via intramuscular injection followed by electroporation at 0, 4th, 8th, 12th week, followed by a 24-week follow-up period. The 5th administration (booster injection) will be conducted at 36th week and subjects will be followed for another 24 weeks. The primary endpoint is safety evaluation of ICVAX in clinically stable HIV-infected patients under ART. The incident rate of adverse events and abnormal laboratory results will be recorded for safety evaluation. The secondary endpoint is immunogenicity evaluation of ICVAX. Antigen-specific cellular and humoral immune responses induced by ICVAX, as well as the effect of ICVAX-ART combined treatment on the viral reservoir, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Tested positive for HIV-1 infection;
2. Aged 18-50, both male and female;
3. Received ART treatment for ≥ 12 months with no occurrence of drug resistance during the treatment period
4. Had <50 copies/ml of plasma HIV RNA for at least (≥) 12 months prior to screening visit;
5. Had ≥350 cells/μL of CD4+ T cells in the past 6 months and >200 cells/μL of CD4+ T cells at the beginning of ART;
6. Adopted contraception method approved by the investigator from 14 days before the first dose to at least 12 weeks after the last dose;
7. Understands the study and voluntarily sign the ICF

Exclusion Criteria:

1. Women who are pregnant or breastfeeding or those who plan to give birth in coming two years (including the subject and his/her spouse);
2. ART has been suspended for more than 2 weeks in the past;
3. Participated in other clinical trials within 24 weeks before the screening visit;
4. Has any opportunistic infections or opportunistic tumors that require systemic treatment within 30 days before being recruited; Has any medical event that the investigator believes will affect the safety and immunogenicity evaluation of the drug;
5. Has a history of autoimmune diseases; a history of severe allergies, such as urticaria, dyspnea, edema, abdominal pain and other symptoms after administration, especially those who have hypersensitivity to the drug components of this study;
6. Received approved vaccines within the past 3 months;
7. Received any blood products, immunoglobulin products, or immunosuppressants within 12 weeks before being recruited;
8. Used interferon, systemic corticosteroids, or other immunosuppressants within the last 3 months (except for local application only);
9. Infected by chronic hepatitis B virus or hepatitis C virus (HBsAg positive or HCV antibody positive)
10. Has any abnormal laboratory results including: neutrophil <1×109/L, serum creatinine>ULN, ALT or AST>1.5×ULN, hemoglobin<80g/L;
11. Has any medical history or clinical manifestations of any physical or mental illness that may affect the subject's completion of this study;
12. Sensitive population to stimulation induced by electrical pulses；Implanted with pacemaker or Automatic Implantable Cardioverter Defibrillator (AICD)
13. Needle phobia
14. Has contraindications for intramuscular administration such as confirmed thrombocytopenia, any coagulation dysfunction or being receiving anticoagulation therapy
15. The investigator considers that he/she is not suitable to participate in this trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events at week 36 [Safety and Tolerability] | Week 36
  The incidence of adverse events and abnormal laboratory results are recorded for safety evaluation at week 36.

SECONDARY OUTCOMES:
Incidence of adverse events at week 60 [Safety and Tolerability] | Week 60
  The incidence of adverse events and abnormal laboratory results are recorded for safety evaluation at week 60.
Antigen-specific T cell responses induced by ICVAX [Immunogenicity] | Week 60
  Antigen-specific T cell responses induced by ICVAX are assessed at week 60 via EliSpot.
Antigen-specific binding antibody responses induced by ICVAX [Immunogenicity] | Week 60
  Antigen-specific binding antibody responses induced by ICVAX are assessed at week 60 via ELISA.
The effect of ICVAX-ART combined treatment on the viral reservoir of HIV-infected patients | Week 60
  The effect of ICVAX-ART combined treatment on the viral reservoir of HIV-infected patients is evaluated at week 60 via PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, Master of Medicine, Principal Investigator — Shenzhen Third People's Hospital; Hongzhou Lu, Doctor of Medicine, Principal Investigator — Shenzhen Third People's Hospital
Locations (1):
- Shenzhen Third People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The results of this study will be publicly disseminated by ways of publication(s) in peer-reviewed scientific journal(s), presentation(s) in scientific conference(s), posting on public clinical trial registry(ies) and/or otherwise instead of individual participant data (IPD) sharing.